CLINICAL TRIAL: NCT05026476
Title: Evaluation of the Acceptability (including Gastrointestinal Tolerance, Compliance) of a Thickener
Brief Title: Acceptability and Tolerance Study of a Thickener
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: RJ1
Record Dates: First submitted 2021-08-24; First posted 2021-08-30 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Dietary Supplement: Resource Thicken up Junior — Each infant and child will be switch over to receive for a period of 7 days (new thickener)

SUMMARY:
This is a prospective, acceptability study to evaluate the gastrointestinal tolerance and compliance of a thickener for the management of reflux, GORD and dysphagia

DETAILED DESCRIPTION:
To evaluate the gastrointestinal tolerance and compliance of a thickener for 7 days for the submission to the Advisory Committee for Borderline Substances (ACBS).

ELIGIBILITY:
Inclusion Criteria:

I. Infants and children aged 6 months and over who require a thickener for reflux, GORD, dysphagia II. Infants and children already on a thickener for the management of reflux, GORD and dysphagia III. Parents to avoid introducing new weaning/ new foods (for the older infants) whilst on the thickener for 1 week when measuring GI tolerance and thickener intake IV. Willingly given, written, informed consent from patient or parent/guardian

Exclusion Criteria:

I. Inability to comply with the study protocol, in the opinion of the investigator.

II. Contraindications to any feed ingredients (see nutritional table and ingredients list) III. Allergy to milk (thickener is made in a factory that handles milk) IV. Children under the age of 6 months of age V. Emergencies VI. Participation in another interventional study

-

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: infants and children
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal tolerance | 7 days
  Measure using daily diary

SECONDARY OUTCOMES:
Participant compliance | 7 days
  Daily intake using diary

CONTACTS AND LOCATIONS:
Overall Officials: Analou Sugar, Principal Investigator — Chelsea and Westminster
Locations (1):
- Chelsea and Westminster Hospital Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No